CLINICAL TRIAL: NCT00869310
Title: Aprepitant in the Prevention of Cisplatin-induced Delayed Emesis: a Double-blind Randomized Trial
Brief Title: Aprepitant in the Prevention of Cisplatin-induced Delayed Emesis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: we terminated the study before enrolling 303/560 due to a slow accrual
Sponsor: S. Maria Hospital, Terni (Other)
Responsible Party: Principal Investigator, Roila Fausto, Dr, S. Maria Hospital, Terni
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IGAR-01-2009; 2008-001339-37
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Emesis
Keywords: aprepitant; delayed emesis; cisplatin; antiemetic
MeSH Terms: conditions — Vomiting | interventions — Aprepitant; Dexamethasone; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Dexamethasone plus Aprepitant
  Interventions: Drug: aprepitant + dexamethasone
- 2 (Active Comparator): dexamethasone plus metoclopramide
  Interventions: Drug: metoclopramide + dexamethasone

INTERVENTIONS:
Drug: aprepitant + dexamethasone — Dexamethasone 8 mg orally: 24 hours after chemotherapy (day 2) and then at 8 am on days 3-4 plus Aprepitant 80 mg orally: 24 hours after chemotherapy on day 2 and then at 8 am on day 3.
  Arms: 1
Drug: metoclopramide + dexamethasone — dexamethasone 8 mg orally: 24 hours after chemotherapy and at 8 pm on day 2, then at 8 am and 8 pm on days 3-4 plus Metoclopramide 20 mg orally 4 times a day: 24 hours after chemotherapy and then at 4 pm, 7 pm, 10 pm on day 2 then at 7 am, 12 am, 5 pm, 10 pm on days 3-4.
  Arms: 2

SUMMARY:
The aim of the study is to compare efficacy and tolerability of aprepitant plus dexamethasone versus metoclopramide plus dexamethasone in the prevention of cisplatin-induced delayed emesis in patients that received aprepitant, palonosetron and dexamethasone before chemotherapy administration for the prevention of acute emesis.

DETAILED DESCRIPTION:
This is a phase III, double-blind, randomized trial, to evaluated the efficacy and safety of aprepitant for the prevention of delayed emesis in patients submitted for the first time to chemotherapy with cisplatin.

The study will be carried out during the first cycle of chemotherapy.

For the prevention of acute emesis, all patients will receive, before chemotherapy:

* dexamethasone 12 mg iv, in 15 minutes, 30 minutes before chemotherapy
* palonosetron 0.25 mg iv bolus, 30 minutes before chemotherapy
* aprepitant 125 mg orally, 60 minutes before chemotherapy

After 24 hours from chemotherapy administration, patients will be randomized to receive one of the following antiemetic treatments:

A) dexamethasone 8 mg orally: 24 hours after chemotherapy and at 8 pm on day 2, then at 8 am and 8 pm on days 3-4 plus Metoclopramide 20 mg orally 4 times a day: 24 hours after chemotherapy and then at 4 pm, 7 pm, 10 pm on day 2 then at 7 am, 12 am, 5 pm, 10 pm on days 3-4.

B) Dexamethasone 8 mg orally: 24 hours after chemotherapy (day 2) and then at 8 am on days 3-4 plus Aprepitant 80 mg orally: 24 hours after chemotherapy on day 2 and then at 8 am on day 3.

The patients will receive prochlorperazine suppositories as rescue medication, for important nausea and vomiting (> 2 episodes) during days 1-5 after chemotherapy.

The patients will receive a diary, which includes a Visual Analogue Scale (VAS) for nausea and vomiting evaluation. All patients will fill out the diary, in which, for 6 consecutive days (days 1-6), patients will report for each day the number of vomiting episodes, the intensity and duration of nausea, any antiemetic rescue medication and any adverse event and its treatment.

In addition, on day 1 before chemotherapy and then on day 6, patients have to fill out the FLIE (Functional Living Index-Emesis), a questionnaire concerning the impact of nausea and vomiting on their quality of life.

Primary end-point is the percentage of complete responses (no vomiting and no rescue treatment) on days 2-5 after cisplatin administration

ELIGIBILITY:
Inclusion Criteria:

1. patients receiving for the first time chemotherapy with cisplatin at doses ≥50 mg/m2.
2. patients over 18 years old and those who signed informed consent
3. adequate contraception if premenopausal women.

Every other anticancer drug in the first 24 hours will be administered after the end of cisplatin.

Exclusion Criteria:

1. patients receiving other anticancer drugs on days 2-4, except 5-fluorouracil, VP16, VM26, vincristine, vinblastine, vindesine, vinorelbine, gemcitabine
2. patients already submitted to chemotherapy with cisplatin
3. patients with concomitant severe diseases, other than neoplasm, or with predisposition to emesis such as intestinal obstruction, active peptic ulcer, hypercalcemia and brain metastases
4. contraindications to corticosteroids (i.e., active peptic ulcer or previous bleeding from peptic ulcer
5. patients submitted to concomitant radiotherapy or submitted to radiotherapy in the 15 days before chemotherapy or planned to receive radiotherapy during the 8 days after chemotherapy
6. patients receiving other concomitant antiemetic treatments or submitted to antiemetic treatments in the 24 hours before chemotherapy
7. patients with nausea or vomiting in the 24 hours before chemotherapy
8. patients receiving concomitant steroids, except when administered at physiologic dose
9. patients receiving concomitant benzodiazepines, except when used for nocturnal sedation
10. patients with WBC count <3000/mm3 or platelet count <70000/mm3
11. patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2009-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Percentage of complete responses (no vomiting and no rescue treatment) on days 2-5 after cisplatin administration | 6 days

SECONDARY OUTCOMES:
Evaluation of the impact on quality of life of the two antiemetic regimens | 6 days
Evaluation of the prognostic factors of delayed emesis in patients receiving a combination of aprepitant, palonosetron, dexamethasone for the prevention of acute emesis | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Roila, MD, Principal Investigator — Oncology Division, S. Maria Hospital, Terni, Italy
Locations (1):
- Fausto Roila, Terni, Terni, Italy

REFERENCES:
- [Result] Hesketh PJ. Potential role of the NK1 receptor antagonists in chemotherapy-induced nausea and vomiting. Support Care Cancer. 2001 Jul;9(5):350-4. doi: 10.1007/s005200000199. PMID 11497388
- [Result] Poli-Bigelli S, Rodrigues-Pereira J, Carides AD, Julie Ma G, Eldridge K, Hipple A, Evans JK, Horgan KJ, Lawson F; Aprepitant Protocol 054 Study Group. Addition of the neurokinin 1 receptor antagonist aprepitant to standard antiemetic therapy improves control of chemotherapy-induced nausea and vomiting. Results from a randomized, double-blind, placebo-controlled trial in Latin America. Cancer. 2003 Jun 15;97(12):3090-8. doi: 10.1002/cncr.11433. PMID 12784346
- [Result] Hesketh PJ, Grunberg SM, Gralla RJ, Warr DG, Roila F, de Wit R, Chawla SP, Carides AD, Ianus J, Elmer ME, Evans JK, Beck K, Reines S, Horgan KJ; Aprepitant Protocol 052 Study Group. The oral neurokinin-1 antagonist aprepitant for the prevention of chemotherapy-induced nausea and vomiting: a multinational, randomized, double-blind, placebo-controlled trial in patients receiving high-dose cisplatin--the Aprepitant Protocol 052 Study Group. J Clin Oncol. 2003 Nov 15;21(22):4112-9. doi: 10.1200/JCO.2003.01.095. Epub 2003 Oct 14. PMID 14559886
- [Result] Roila F, Hesketh PJ, Herrstedt J; Antiemetic Subcommitte of the Multinational Association of Supportive Care in Cancer. Prevention of chemotherapy- and radiotherapy-induced emesis: results of the 2004 Perugia International Antiemetic Consensus Conference. Ann Oncol. 2006 Jan;17(1):20-8. doi: 10.1093/annonc/mdj078. Epub 2005 Nov 28. PMID 16314401
- [Result] Chawla SP, Grunberg SM, Gralla RJ, Hesketh PJ, Rittenberg C, Elmer ME, Schmidt C, Taylor A, Carides AD, Evans JK, Horgan KJ. Establishing the dose of the oral NK1 antagonist aprepitant for the prevention of chemotherapy-induced nausea and vomiting. Cancer. 2003 May 1;97(9):2290-300. doi: 10.1002/cncr.11320. PMID 12712486
- [Result] Aapro MS, Grunberg SM, Manikhas GM, Olivares G, Suarez T, Tjulandin SA, Bertoli LF, Yunus F, Morrica B, Lordick F, Macciocchi A. A phase III, double-blind, randomized trial of palonosetron compared with ondansetron in preventing chemotherapy-induced nausea and vomiting following highly emetogenic chemotherapy. Ann Oncol. 2006 Sep;17(9):1441-9. doi: 10.1093/annonc/mdl137. Epub 2006 Jun 9. PMID 16766588
- [Result] Ondansetron versus metoclopramide, both combined with dexamethasone, in the prevention of cisplatin-induced delayed emesis. The Italian Group for Antiemetic Research. J Clin Oncol. 1997 Jan;15(1):124-30. doi: 10.1200/JCO.1997.15.1.124. PMID 8996133
- [Derived] Roila F, Ruggeri B, Ballatori E, Fatigoni S, Caserta C, Licitra L, Mirabile A, Ionta MT, Massidda B, Cavanna L, Palladino MA, Tocci A, Fava S, Colantonio I, Angelelli L, Ciuffreda L, Fasola G, Zerilli F. Aprepitant versus metoclopramide, both combined with dexamethasone, for the prevention of cisplatin-induced delayed emesis: a randomized, double-blind study. Ann Oncol. 2015 Jun;26(6):1248-1253. doi: 10.1093/annonc/mdv132. Epub 2015 Mar 5. PMID 25743855